CLINICAL TRIAL: NCT06136221
Title: Testing LiverWatch, a Home-Based Remote-Monitoring Intervention for Advanced Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 844700
Record Dates: First submitted 2023-10-30; First posted 2023-11-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cirrhosis, Liver; End Stage Liver DIsease; Symptoms and Signs; Physical Inactivity; Muscle Loss
Keywords: Telehealth; Remote Symptom Monitoring; Gamification
MeSH Terms: conditions — Liver Cirrhosis; End Stage Liver Disease; Signs and Symptoms; Sedentary Behavior; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: This is a longitudinal intervention study utilizing diverse cohorts of patients with cirrhosis. It is a 2-arm, patient-randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (No Intervention): Patients will undergo baseline interviews with study coordinators. All participants will be screened for malnutrition with the validated malnutrition screening tool (MST). At the baseline interview, patients will receive instructional handouts on dietary changes and recipes as per the updated 2019 European Society for Clinical Nutrition & Metabolism (ESPEN) guidelines. Information on the resource CirrhosisCare.ca will also be provided. Participants in the control arm will receive Fitbits to monitor their steps. They will be asked to try and get up to 7000 steps per day, and no follow-up on their progress in terms of step counts will be given during the 12 weeks. All participants will be allowed to keep their Fitbit once they complete the study.
- LiverWatch Intervention (Experimental): Patients will undergo symptom-based monitoring with targeted nutrition support. participants in Arm 2 will also receive educational text messages related to cirrhosis and physical activity. In summary, there are four components to the
  * Remote Symptom Monitoring
  * Targeted Nutrition Assessment and Intervention
  * Physical Activity and Rewards Program
  * Motivational Messages
  Subjects will be enrolled in an online portal, Way to Health (W2H), which automates many of the research and monitoring functions of the intervention. Patients will receive remote symptom monitoring on a weekly basis, enhanced nutrition assistance through weekly education videos, and "motivational messages" on Mondays and Fridays that include education on diet, physical activity, and cirrhosis. Participants in this arm will also be encouraged to increase their step count using a rewards system built through the W2H.
  Interventions: Behavioral: LiverWatch Intervention

INTERVENTIONS:
Behavioral: LiverWatch Intervention — The LiverWatch Intervention will include standard cirrhosis care and include additional components utilizing the W2H system. Details on this intervention are included in the study arm description.
  Arms: LiverWatch Intervention

SUMMARY:
Remote healthcare monitoring for cirrhosis has shown promise in overcoming barriers to accessing specialty care, improving healthcare quality, and reducing mortality. The LiverWatch study is investigating whether a remote nutrition, physical activity, and education intervention can improve health outcomes in those with cirrhosis. In this clinical trial, individuals will be randomized to either enhanced usual care or the LiverWatch intervention. Both groups are given fitbits and asked to increase their step counts. Those in the Liverwatch group will be incentivized for increase their physical activity while also undergoing a personalized nutrition intervention and weekly symptom monitoring and cirrhosis education.

DETAILED DESCRIPTION:
Liver cirrhosis is a chronic condition with a high symptom burden, morbidity, mortality and costs. Common symptoms and reasons for hospitalizations in cirrhosis are 'fluid overload' (e.g. abdominal and leg swelling), hepatic encephalopathy (episodic cognitive impairment), physical frailty, and infections. Pilot and feasibility data show that many of these complications may be managed remotely with patient and caregiver-directed text-messaging platforms, online portals, and frequent telephone check-ins with the clinical team. This approach can help reduce unnecessary urgent visits and hospitalizations. Malnutrition is present among an estimated 60% of patients with advanced cirrhosis, and is associated with frailty, loss of muscle mass, and hepatic encephalopathy, leading to a greater likelihood of hospitalization and poorer health-related quality of life (HRQoL). Studies show that HRQoL may improve with targeted nutritional management, yet personalized nutritional interventions are not routinely incorporated into many telehealth and remote monitoring approaches for cirrhosis. To be effective, telehealth and remote monitoring interventions must be patient-centered, feasible, acceptable, and sustainable.

The LiverWatch study is investigating whether an intervention aimed at improving physical health and wellness as well as monitor for symptoms in those with cirrhosis is an effective strategy to improve patient-centered outcomes. This study compares enhanced usual care of those with cirrhosis versus an intervention that includes a dietitian consultation, educational messages, and a step rewards program. LiverWatch leverages the use of electronic health records and Way To Health (W2H) text messages to explore its aims. LiverWatch is a 2-arm, patient-randomized controlled trial at the University of Pennsylvania. A total of 110 patients with cirrhosis aged 18 or older (n=55 per arm) will be recruited and randomized to intervention versus enhanced usual care for 12 weeks with a 12 week follow-up period. Study visits will occur at Baseline (Week 0), Week 6, and Week 12. Clinical outcomes will be measured from the electronic medical record (EMR) at Week 24. The LiverWatch intervention includes:

* Modifiable walking goals with the use of W2H and a fitbit.
* Cirrhosis, nutrition, and fitness education sent weekly via text message
* A one-one baseline visit with a registered dietitian to discuss healthy eating habits and set up individualized goals
* Remote symptom monitoring conducted via text message

The primary objective of the study is to test the effectiveness of LiverWatch. The secondary objective is to explore barriers to and facilitators of optimal implementation and scalability of LiverWatch among patients, caregivers, clinicians, and health-system administrators.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Aged 18 years or older
* Home-dwelling
* Diagnosis of cirrhosis- Child Turcotte-Pugh (CTP) B or C or a complication in the past 6 months (CTP B or higher, hepatic encephalopathy, variceal bleeding, fluid overload, liver-related hospitalization, or requiring symptom management with diuretics, non-absorbable disaccharides, rifaximin, nonselective beta blockers)
* Patient and/or caregiver is able and willing to receive SMS text messages
* Willing and able to wear personal fitness trackers and engage with study staff

Exclusion Criteria:

* No access to a smartphone
* Non-home dwelling
* On hospice care
* Model for end stage liver disease (MELD) score ≥30
* Advanced hepatocellular carcinoma, BCLC C or higher
* Hospitalization within the last 30 days
* Deemed not appropriate by treating physician for medical reasons
* Enrolled in other dietary or physical activity interventions
* Receiving physical therapy as standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS 29+2 | 12 Weeks
  The PROMIS 29+2 assessment measures seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance). There are four questions asked for each of the domains along with the two questions pertaining to cognition. These domains are measured on a Likert scale (units: 1-5) and are universal regardless of disease state.

SECONDARY OUTCOMES:
Automated Self-Administered 24-hour Dietary Assessment Tool | 12 Weeks
  The Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool is a free, web-based application that enables multiple, automatically coded, self-administered 24-hour diet recalls and/or food diaries. The ASA24 consists of two websites. The ASA24 respondent website guides participants through the completion of either 24-hour recalls or food records. The calories consumed from these meals will be measured.
Average Daily Step Count | 12 Weeks
  The average daily step count will be measured in both groups longitudinally over 12 weeks using Fitbit.
MoCA for the Blind | 12 Weeks
  We will assess global cognition with the Montreal Cognitive Assessment (MoCA), a well-validated cognitive assessment used in diverse clinical settings and validated in liver disease. The MoCA for the Blind version can be administered remotely over the phone to participants. Participant performance is measured on a scale of 0-30.
Simplified Animal Naming Test (S-ANT) | 12 Weeks
  The Simplified Animal Naming Test (S-ANT) is a cognitive assessment used to assess semantic fluency that becomes impaired in hepatic encephalopathy. Participants have 60 seconds to name as many animals as they can without repeating names. The number of animals named by participants during this time frame will be counted.
Grip Strength | 12 Weeks
  Grip strength is assessed using the participant's dominant hand with the Jamar+® Digital Dynamometer. Units are in lbs., and an average of 3 age- and sex-adjusted measures is calculated.
Balance | 12 Weeks
  Balance is assessed with the participant performing three different stances (feet side-by-side, semi-tandem, and tandem). The length of time a participant is able to maintain these stances is measured in seconds, up to 10 seconds for each stance.
30-Second Chair Test | 12 Weeks
  The 30-Second Chair Stand test is a measure of leg strength and endurance. The patient is asked to move from a seated position with arms crossed over the into the standing position and then sit back down. The test administrator counts the number of times the patient comes to a full standing position in 30 seconds. The number of successful completions indicates the risk of fall.
Days Alive and Out of Hospital (DAOH) | 24 Weeks
  The number of days a patient spends alive and not hospitalized for any reason.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania